CLINICAL TRIAL: NCT02126189
Title: An Epidemiological Study of Mucosal Squamous Cell Carcinomas of the Head and Neck
Brief Title: The Princess Alexandra Hospital and the QIMR Berghofer Medical Research Institute Head and Neck Cancer Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Queensland Centre of Excellence for Head and Neck Cancer (Other)
Collaborators: QIMR Berghofer Medical Research Institute (Other); Princess Alexandra Hospital, Brisbane, Australia (Other); Translational Research Institute, Brisbane, Australia (Unknown); The University of Queensland (Other)
Responsible Party: Sponsor
Other Study IDs: HREC13QPAH36
Record Dates: First submitted 2014-04-23; First posted 2014-04-29 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Human Papillomavirus
Keywords: Head and Neck Squamous Cell Carcinoma; Human Papillomavirus; Aetiology; prevalence; risk factors; clinical outcome
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Case-Control
Biospecimen Retention: Samples With DNA — Participants are asked to give their consent for researchers to obtain tissue from tumour blocks. This tissue is taken as part of their normal care and treatment. If consent is given, formalin-fixed paraffin embedded (FFPE) tissue samples will be used to determine HPV status.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Head and neck cancer: All patients presenting to the Head and Neck Cancer Clinic at the Princess Alexandra Hospital, Brisbane, Australia are invited to participate.

SUMMARY:
This study is designed to refine the aetiological causes of cancers of the head and neck and investigate the ways in which human papillomavirus and life-style factors cause head and neck cancers. This study will determine if these factors affect the treatment of cancer.

All patients attending the Head and Neck Clinic at the Princess Alexandra Hospital is invited to complete a risk factor questionnaire and give consent for their clinical data and tissue samples to be available for future research activities. The risk factor questionnaire is based on existing validated instruments developed by the QIMR Berghofer Medical Research Institute Cancer Control Group, and will collect standardised information relating to demographics and causal factors (tobacco and alcohol intake), risk modifiers (dentition, asprin and non-steroidal anti-inflammatory drugs (NSAIDS), height, weight, physical activity, diet quality etc) and behaviours (oral sex etc)

DETAILED DESCRIPTION:
Data is collected using a simple four-page paper-based questionnaire. Information to be collected include age, sex, height and weight (at age 20, current age, and heaviest ever), history of cancer (own and partner). Questions about recreational physical activity, smoking history and alcohol consumption, acid reflux, heartburn, denture use and tonsillectomy, frequency of use of paracetamol, antihistamine and NSAIDS.

The questionnaires also ask participants some detailed questions about sexual behaviour and history if they are comfortable to give this information.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting to the Head and Neck Cancer Clinic at the Princess Alexandra Hospital Brisbane Australia.

Exclusion Criteria:

* nil

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients presenting to the Head and Neck Cancer Clinic at the Princess Alexandra Hospital, Brisbane, Australia. Patients may be be new patients or old patients and may have a new diagnosis or they may have a recurrence.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2013-11; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
To identify exposures associated with an increased risk of head and neck squamous cell carcinoma | 2 years

OTHER OUTCOMES:
To compare subjects who have ever been exposed with those who have never been exposed. | 2 years
To estimate the effect of each exposure adjusted for the confounding effects of other exposures. | 2 years
To test for trends in head and neck squamous cell carcinoma | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Annika Antonsson, Dr, Principal Investigator — QIMR Berghofer Medical Research Institute; Ben Panizza, Assoc Prof, Principal Investigator — Princess Alexandra Hospital; Sandro Porceddu, Assoc Prof, Principal Investigator — Princess Alexandra Hospital; David Whiteman, Prof, Principal Investigator — QIMR Berghofer Medical Research Institute
Locations (1):
- Princess Alexandra Hospital, Brisbane, Queensland, Australia